CLINICAL TRIAL: NCT01448954
Title: A Randomised, Placebo-Controlled, Double-Blind, Parallel Group Phase II Study to Assess the Safety, Tolerability and Pharmacokinetics of ADC3680B in Subjects With Partly Controlled Atopic Asthma
Brief Title: A Study to Evaluate Safety, Tolerability and Pharmacokinetics of ADC3680B in Subjects With Partly Controlled Atopic Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pulmagen Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADC3680-04
Record Dates: First submitted 2011-09-26; First posted 2011-10-07 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Atopic Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADC3680B oral (Experimental)
  Interventions: Drug: ADC3680B oral
- Placebo oral (Placebo Comparator)
  Interventions: Drug: Placebo oral

INTERVENTIONS:
Drug: ADC3680B oral — Once daily for 28 days
  Arms: ADC3680B oral
Drug: Placebo oral — Once daily for 28 days
  Arms: Placebo oral

SUMMARY:
This study is to examine the safety, tolerability, pharmacokinetics and functional activity of ADC3680B administered once daily for 28 days in subjects with partly controlled atopic asthma.

ELIGIBILITY:
Inclusion Criteria:

* Partially controlled mild-moderate atopic asthma
* Receiving inhaled corticosteroids
* Non-smoker or former smoker
* Males and females aged 18 to 55 years inclusive
* If female, must be of non-childbearing potential

Exclusion Criteria:

* History of acute severe asthma attacks
* History of COPD
* Other serious respiratory or other medical condition which may interfere with the outcome of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of the change in frequency and severity of adverse events as a measure of safety and tolerability | Baseline to Day 35
Evaluation of the change in incidence of routine haematology and biochemistry abnormalities as a measure of safety | Baseline to Day 35
Evaluation of the change in vital signs as a measure of safety | Baseline to Day 35
Evaluation of the change in Pulmonary function as a measure of safety and tolerability | Baseline to Day 35
Assessment of the change in asthma symptoms using the Asthma Control Questionnaire as a measure of safety and tolerability | Baseline to Day 28

SECONDARY OUTCOMES:
Determination of concentrations of ADC3680B in plasma | Days 1-2 and Days 28-30
Exploratory assessment of exhaled nitric oxide and selected markers of inflammation in blood | Day 1 and Day 28

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Belfast
  - Manchester